





Enjoy Your Bump v3.0. 5th July 2017

## CONSENT FORM - Enjoy Your Bump

## Feasibility Study Investigating the Acceptableness and Efficacy of a Pregnancy Focussed Online Cognitive Behavioural Therapy Package

| Participant ID: | | | | | |
|---|---|---|---|---|---|
| Prof Rebecca Reynolds, Clinical Reader & Honorary Consultant, University of Edinburgh Dr Fiona Denison, Consultant Obstetrician, University of Edinburgh | | | | | |
| | | | | Please i | nitial box |
| 1. | I confirm that I have read and understand the information sheet (as specified in this document header) for the above study and have had the opportunity to consider the information and ask questions. | | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | | | |
| 3. | , | | | | |
| | may be looked at by members of the study team, individuals from the Sponsor, from the NHS organisation or other authorities, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | | L |
| 4. | I agree to my General Practitioner being informed of my participation in this study. | | | | |
| 5. | Lundaretand that the 'Enjay Vour Pump' website is owned by a company (Five Areas Ltd) | | | | |
| J. | I understand that the 'Enjoy Your Bump' website is owned by a company (Five Areas Ltd) who are independent of NHS Lothian and the University of Edinburgh. I am aware that I will | | | | |
| | be given the opportunity to read and decide whether to accept their Terms and Conditions and Privacy Policy before registering my details on the website. | | | | |
| 6. | 6. I agree to take part in the above study. | | | | |
| Name of Participant | | Date | Signature | | |
| Name of Person taking consent | | Date | Signature | | |

1x original – into Site File; 1x copy – to Participant; 1x copy – into medical records